CLINICAL TRIAL: NCT00805441
Title: A Phase 2 Study of LY686017 Compared With Placebo for the Treatment of Alcohol Dependence
Brief Title: A Study in the Treatment of Alcohol Dependence.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12422; H8R-MC-HJAQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Dependence
Keywords: Alcoholic
MeSH Terms: conditions — Alcoholism | interventions — LY686017

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- LY686017 (Experimental)
  Interventions: Drug: LY686017

INTERVENTIONS:
Drug: LY686017 — 50 milligrams (mg) daily by oral route for 12 weeks
  Arms: LY686017
Drug: Placebo — Daily by oral route for 12 weeks
  Arms: Placebo

SUMMARY:
H8R-MC-HJAQ is a Phase 2, parallel, double-blind, randomized study comparing LY686017 with placebo in a 12-week trial that includes Medical Management. This study is an outpatient study in which approximately 180 alcohol dependent subjects will be enrolled. Subjects will be randomized in a 1:1 fashion to LY686017 or placebo, and will receive once daily dosing for twelve weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have Alcohol Dependence.
* Are men or women who are ambulatory outpatients between 21 to 65 years of age (inclusive) showing evidence of living in a non-custodial stable residence and with no plans to move during the next 5 months.
* Females of childbearing potential (not surgically sterilized and between menopause) must test negative for pregnancy at the time of enrollment based on a pregnancy test. They must agree to use a reliable method of birth control during the study and for 2 months following the last dose of study drug.
* Drink on average more than 14 drinks (women) or 21 drinks (men) per week with at least 2 heavy drinking days per week.
* Endorse abstinence or reduction in drinking as an interim goal toward abstinence.

Exclusion Criteria:

* Are investigator site personnel directly affiliated with this study and/or their immediate families.
* Are Lilly employees.
* Are currently enrolled in or discontinued within the last 30 days from a clinical trial.
* Have experienced an acute alcohol withdrawal syndrome within the past 6 months or are currently or during this study at significant risk of suffering an acute alcohol withdrawal syndrome.
* Have a history of serious head injury, neoplasm or hemorrhage, prior seizure (other than a history of childhood febrile seizure), or other condition that would place the subject at increased risk for seizures.
* Are taking or have taken anticonvulsant medications for seizures.
* Are diagnosed with substance dependence or substance abuse other than alcohol, cannabis, nicotine, or caffeine within 12 months prior to first visit.
* Are receiving medications or intensive behavioral or psychological therapy delivered by a licensed or certified alcohol treatment specialist for alcohol dependence.
* Have signs and symptoms or an active illness within the past 2 weeks of first visit that meet criteria diagnosis of Major Depressive Disorder. In addition, meet criteria as diagnosis for any comorbid Axis I disorders (such as anxiety disorders, obsessive compulsive disorder (OCD), Posttraumatic stress disorder (PTSD), panic disorder, or dysthymia).
* Have a positive urine drug screen for any non-prescribed substances of abuse.
* Have a serious medical illness including but not limited to any cardiovascular, hepatic, respiratory, hematological, endocrine, or neurological disease, or any clinically significant laboratory abnormality.
* Ever had electroconvulsive therapy (ECT).
* Have abnormal thyroid stimulating hormone (TSH) concentrations or are taking thyroid supplements.
* Have a history of cirrhosis or laboratory evidence of hepatocellular injury.
* An abnormality in serum Prothrombin time.
* Are unable to make themselves available for the duration of the study or abide by study procedures and restrictions.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oceanside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Deerfield Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Naperville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Canton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Havertown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeSoto, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlottesville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kirkland, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY686017 | Placebo
Started | 94 | 96
Full Analysis Set (FAS) | 92 (All randomized participants who received ≥1 dose study drug and contributed to post-baseline data.) | 91 (All randomized participants who received ≥1 dose study drug and contributed to post-baseline data.)
Completed | 60 | 60
Not Completed | 34 | 36
Not completed — Adverse Event | 5 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 4 | 8
Not completed — Lost to Follow-up | 10 | 13
Not completed — Withdrawal by Subject | 15 | 9
Not completed — Physician Decision | 0 | 1
Not completed — Acute Alcohol Withdrawal | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all randomized participants who received ≥1 dose study drug and contributed to post-baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY686017 | Placebo | Total
Number analyzed (Participants) | 92 | 91 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (10.5) | 43.0 (11.1) | 43.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 59 | 55 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 86 | 87 | 173
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 21 | 39
  White | 69 | 67 | 136
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 92 | 91 | 183

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Heavy Drinking Days
Description: The Alcohol Timeline Followback (TLFB) is used in calculating the percent reduction in heavy drinking days. The TLFB is a method for assessing the quantity of alcohol consumption on a daily basis. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome. Recorded is the number of standard drinks that have been consumed each day during last 4 weeks. One standard drink on the TLFB was defined as: 12 ounce (oz) beer [5% alcohol by volume (abv)], 5 oz of wine (10-12% abv), 3 oz of fortified wine (16-18% abv), or 1-1.2 oz of hard liquor (86-100 proof; 43-50% abv). Heavy drinking is defined as ≥4 drinks per day for women and ≥5 drinks per day for men.
Time Frame: Baseline, Weeks 4 and 8 and 12 and 16
Population: All randomized participants who received at least one dose of study drug and had daily drinking assessed at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: percent of heavy drinking days
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 91 | 90
percent of heavy drinking days
  Week 4 | -45.63 (36.58) | -39.72 (36.52)
  Week 8: number analyzed (Participants) | 75 | 73
  Week 8 | -60.98 (39.25) | -49.88 (48.43)
  Week 12: number analyzed (Participants) | 65 | 64
  Week 12 | -68.56 (40.01) | -57.44 (42.02)
  Week 16: number analyzed (Participants) | 61 | 61
  Week 16 | -69.46 (35.84) | -59.12 (40.42)

2. Secondary Outcome: Percent Days Abstinent Per Month
Description: The Alcohol Timeline Followback (TLFB) is used in calculating the percentage of days abstinent (days where no alcoholic drinks were consumed). The TLFB is a method for assessing the quantity of alcohol consumption on a daily basis. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome. Recorded is the number of standard drinks that have been consumed each day. One standard drink on the TLFB was defined as: 12 ounce (oz) beer [5% alcohol by volume (abv)], 5 oz of wine (10-12% abv), 3 oz of fortified wine (16-18% abv), or 1-1.2 oz of hard liquor (86-100 proof; 43-50% abv). Percentage days per month= (number of days where no alcoholic beverages were consumed/number of days in a month)*100.
Time Frame: Baseline and Weeks 4 and 8 and 12 and 16.
Population: All randomized participants who received at least one dose of study drug and had daily drinking assessed at the specified time points.
Measure: Mean (Standard Deviation); unit: percentage days abstinent per month
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 92 | 91
percentage days abstinent per month
  Baseline | 11.63 (12.55) | 14.54 (17.32)
  Week 4: number analyzed (Participants) | 91 | 90
  Week 4 | 30.28 (28.13) | 29.44 (26.56)
  Week 8: number analyzed (Participants) | 75 | 73
  Week 8 | 40.73 (32.97) | 40.07 (33.68)
  Week 12: number analyzed (Participants) | 65 | 64
  Week 12 | 51.43 (32.59) | 45.81 (34.74)
  Week 16: number analyzed (Participants) | 61 | 61
  Week 16 | 52.92 (32.07) | 44.63 (36.84)

3. Secondary Outcome: Number of Drinks Per Drinking Day During a Month
Description: The Alcohol Timeline Followback (TLFB) is used in calculating the number of drinks per drinking day. The TLFB is a method for assessing the quantity of alcohol consumption on a daily basis. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome. Recorded is the number of standard drinks that have been consumed each day. One standard drink on the TLFB was defined as: 12 ounce (oz) beer [5% alcohol by volume (abv)], 5 oz of wine (10-12% abv), 3 oz of fortified wine (16-18% abv), or 1-1.2 oz of hard liquor (86-100 proof; 43-50% abv).
Time Frame: Baseline and Weeks 4 and 8 and12 and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: drinks/drinking day/month
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 92 | 91
drinks/drinking day/month
  Baseline | 7.04 (3.07) | 7.35 (3.78)
  Week 4: number analyzed (Participants) | 91 | 90
  Week 4 | 3.92 (2.37) | 4.69 (3.64)
  Week 8: number analyzed (Participants) | 75 | 73
  Week 8 | 3.03 (2.52) | 3.36 (3.31)
  Week 12: number analyzed (Participants) | 65 | 64
  Week 12 | 2.32 (2.25) | 2.99 (3.70)
  Week 16: number analyzed (Participants) | 61 | 61
  Week 16 | 2.31 (2.83) | 2.92 (3.38)

4. Secondary Outcome: Time to First Heavy Drinking Day
Description: The Alcohol Timeline Followback (TLFB) is used to assess the time to first heavy drinking day. The TLFB is a method for assessing the quantity of alcohol consumption on a daily basis. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome. Recorded is the number of standard drinks that have been consumed each day. One standard drink on the TLFB was defined as: 12 ounce (oz) beer [5% alcohol by volume (abv)], 5 oz of wine (10-12% abv), 3 oz of fortified wine (16-18% abv), or 1-1.2 oz of hard liquor (86-100 proof; 43-50% abv). Heavy drinking is defined as ≥4 drinks per day for women and ≥5 drinks per day for men. Those who did not drink are considered to be "censored."
Time Frame: Baseline up to Week 12
Population: All randomized participants who received at least one dose of study drug and had daily drinking assessed. The numbers of participants censored are 4 for LY686017 group and 3 for placebo group.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 91 | 90
days | 7.3 (16.8) | 8.0 (22.2)

5. Secondary Outcome: Change From Baseline in Drinker Inventory of Consequences (DrInC) Subscale and Total Scale
Description: DrInC is a self-administered, 50-item questionnaire designed to measure adverse consequences of alcohol abuse in 5 areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal. All items for the DrInC are scored from 0-3 with higher scores indicating worse adverse consequences. Interpersonal subscale (10 items: scores range from 0-30) measures the impact of drinking on the participants' relationships. Physical subscale (8 items: scores range from 0-24) measures adverse physical states resulting from excessive drinking. Social subscale (7 items: scores range from 0-21) measures role fulfillment. Impulsive subscale (12 items: scores range from 0-36) measures sequelae of over drinking. Intrapersonal subscale (8 items: scores range from 0-24) measures subjective perceptions that may not be readily observable by others. Total scores range from 0-150, with higher scores indicating greater severity of symptoms.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had DrInC assessed at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 92 | 91
units on a scale
  Interpersonal | -2.9 (5.5) | -3.9 (6.8)
  Physical | -3.1 (4.0) | -2.3 (4.3)
  Social | -2.0 (3.4) | -2.1 (4.1)
  Impulsive | -2.5 (4.4) | -2.5 (5.8)
  Intrapersonal | -4.2 (6.7) | -3.7 (6.2)
  Total | -16.2 (22.2) | -16.4 (25.5)

6. Secondary Outcome: Change From Baseline in Alcohol Urge Questionnaire (AUQ)
Description: AUQ measures participant's feeling and thoughts about drinking, and uses a 7 point (1-7) Likert scale for each of 8 items (questions). Scores range from 8 (less urge to drink) to 56 (more urge to drink).
Time Frame: Baseline, Weeks 1 and 2 and 3 and 4 and 6 and 8 and 10 and 12
Population: All randomized participants who received at least one dose of study drug and had AUQ assessed at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 91 | 90
units on a scale
  Week 1 | -2.9 (10.2) | -2.9 (8.8)
  Week 2: number analyzed (Participants) | 86 | 83
  Week 2 | -5.0 (11.5) | -3.6 (11.1)
  Week 3: number analyzed (Participants) | 83 | 79
  Week 3 | -5.3 (10.5) | -6.0 (9.6)
  Week 4: number analyzed (Participants) | 79 | 76
  Week 4 | -5.9 (10.9) | -5.9 (10.1)
  Week 6: number analyzed (Participants) | 75 | 73
  Week 6 | -6.4 (11.0) | -8.5 (11.7)
  Week 8: number analyzed (Participants) | 70 | 66
  Week 8 | -5.8 (10.6) | -7.7 (11.8)
  Week 10: number analyzed (Participants) | 65 | 64
  Week 10 | -5.7 (11.0) | -7.7 (12.7)
  Week 12: number analyzed (Participants) | 64 | 62
  Week 12 | -6.3 (10.6) | -9.0 (12.5)

7. Secondary Outcome: Change From Baseline in Penn Alcohol Craving Scale (PACS)
Description: PACS is a 5-item self-administered instrument that measures frequency, intensity, and duration of thoughts about drinking, ability to resist drinking and craving. Each item ranges from 0-6 with 6 indicating worse symptoms.
Time Frame: Baseline, Weeks 1 and 2 and 3 and 4 and 6 and 8 and 10 and 12
Population: All randomized participants who received at least one dose of study drug and had PACS assessed at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 90 | 90
units on a scale
  Frequency: Week 1 | -1.0 (1.4) | -0.6 (1.3)
  Frequency: Week 2: number analyzed (Participants) | 86 | 83
  Frequency: Week 2 | -1.3 (1.4) | -1.0 (1.3)
  Frequency: Week 3: number analyzed (Participants) | 83 | 79
  Frequency: Week 3 | -1.4 (1.5) | -1.0 (1.3)
  Frequency: Week 4: number analyzed (Participants) | 79 | 76
  Frequency: Week 4 | -1.5 (1.6) | -1.3 (1.3)
  Frequency: Week 6: number analyzed (Participants) | 75 | 73
  Frequency: Week 6 | -1.5 (1.6) | -1.3 (1.3)
  Frequency: Week 8: number analyzed (Participants) | 70 | 66
  Frequency: Week 8 | -1.5 (1.5) | -1.3 (1.4)
  Frequency: Week 10: number analyzed (Participants) | 65 | 64
  Frequency: Week 10 | -1.7 (1.6) | -1.3 (1.3)
  Frequency: Week 12: number analyzed (Participants) | 64 | 62
  Frequency: Week 12 | -1.7 (1.5) | -1.4 (1.4)
  Intensity: Week 1 | -1.2 (1.7) | -0.7 (1.4)
  Intensity: Week 2: number analyzed (Participants) | 86 | 83
  Intensity: Week 2 | -1.6 (1.6) | -1.0 (1.3)
  Intensity: Week 3: number analyzed (Participants) | 83 | 79
  Intensity: Week 3 | -1.7 (1.7) | -1.3 (1.4)
  Intensity: Week 4: number analyzed (Participants) | 79 | 76
  Intensity: Week 4 | -1.8 (1.8) | -1.4 (1.6)
  Intensity: Week 6: number analyzed (Participants) | 75 | 73
  Intensity: Week 6 | -2.0 (2.0) | -1.6 (1.7)
  Intensity: Week 8: number analyzed (Participants) | 70 | 66
  Intensity: Week 8 | -2.0 (1.8) | -1.5 (1.7)
  Intensity: Week 10: number analyzed (Participants) | 65 | 64
  Intensity: Week 10 | -2.1 (1.8) | -1.6 (1.6)
  Intensity: Week 12: number analyzed (Participants) | 64 | 62
  Intensity: Week 12 | -2.2 (1.6) | -1.8 (1.7)
  Duration: Week 1 | -0.9 (1.6) | -0.4 (1.6)
  Duration: Week 2: number analyzed (Participants) | 86 | 83
  Duration: Week 2 | -1.1 (1.7) | -0.6 (1.7)
  Duration: Week 3: number analyzed (Participants) | 83 | 79
  Duration: Week 3 | -1.2 (1.8) | -0.7 (1.5)
  Duration: Week 4: number analyzed (Participants) | 79 | 76
  Duration: Week 4 | -1.1 (1.7) | -0.8 (1.5)
  Duration: Week 6: number analyzed (Participants) | 75 | 73
  Duration: Week 6 | -1.3 (1.9) | -0.9 (1.6)
  Duration: Week 8: number analyzed (Participants) | 70 | 66
  Duration: Week 8 | -1.2 (1.6) | -1.0 (1.8)
  Duration: Week 10: number analyzed (Participants) | 65 | 64
  Duration: Week 10 | -1.2 (1.8) | -1.0 (1.6)
  Duration: Week 12: number analyzed (Participants) | 64 | 62
  Duration: Week 12 | -1.4 (1.8) | -1.0 (1.8)
  Resistance: Week 1 | -1.2 (1.6) | -0.9 (1.7)
  Resistance: Week 2: number analyzed (Participants) | 86 | 83
  Resistance: Week 2 | -1.4 (1.7) | -1.0 (1.8)
  Resistance: Week 3: number analyzed (Participants) | 83 | 79
  Resistance: Week 3 | -1.4 (1.8) | -1.2 (1.6)
  Resistance: Week 4: number analyzed (Participants) | 79 | 76
  Resistance: Week 4 | -1.6 (1.9) | -1.3 (1.7)
  Resistance: Week 6: number analyzed (Participants) | 75 | 73
  Resistance: Week 6 | -1.6 (2.0) | -1.5 (2.0)
  Resistance: Week 8: number analyzed (Participants) | 70 | 66
  Resistance: Week 8 | -1.8 (1.9) | -1.5 (1.9)
  Resistance: Week 10: number analyzed (Participants) | 65 | 64
  Resistance: Week 10 | -1.7 (1.9) | -1.5 (1.8)
  Resistance: Week 12: number analyzed (Participants) | 64 | 62
  Resistance: Week 12 | -1.9 (1.8) | -1.4 (1.8)
  Craving: Week 1 | -1.0 (1.2) | -0.6 (1.2)
  Craving: Week 2: number analyzed (Participants) | 86 | 83
  Craving: Week 2 | -1.2 (1.3) | -0.9 (1.2)
  Craving: Week 3: number analyzed (Participants) | 83 | 79
  Craving: Week 3 | -1.4 (1.3) | -1.1 (1.2)
  Craving: Week 4: number analyzed (Participants) | 79 | 76
  Craving: Week 4 | -1.5 (1.4) | -1.2 (1.2)
  Craving: Week 6: number analyzed (Participants) | 75 | 73
  Craving: Week 6 | -1.7 (1.4) | -1.4 (1.3)
  Craving: Week 8: number analyzed (Participants) | 70 | 66
  Craving: Week 8 | -1.7 (1.4) | -1.4 (1.3)
  Craving: Week 10: number analyzed (Participants) | 65 | 64
  Craving: Week 10 | -1.6 (1.4) | -1.4 (1.2)
  Craving: Week 12: number analyzed (Participants) | 64 | 62
  Craving: Week 12 | -1.8 (1.4) | -1.5 (1.3)

8. Secondary Outcome: Change From Baseline in Beck Depression Inventory II (BDI-II) Total Score
Description: BDI-II is a 21-item, participant-completed questionnaire to assess characteristics of depression. There is a 4-point scale for each item ranging from 0 (no depression) to 3 (very depressed). Total scores range from 0-63. Higher scores indicate greater severity of depression.
Time Frame: Baseline, Weeks 1 and 2 and 3 and 4 and 6 and 8 and 10 and 12
Population: All randomized participants who received at least one dose of study drug and had BDI-II assessed at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 91 | 90
units on a scale
  Week 1 | 0.0 (4.1) | -1.4 (3.6)
  Week 2: number analyzed (Participants) | 86 | 83
  Week 2 | -0.9 (4.1) | -1.0 (3.9)
  Week 3: number analyzed (Participants) | 83 | 79
  Week 3 | -1.5 (4.7) | -1.2 (3.9)
  Week 4: number analyzed (Participants) | 79 | 76
  Week 4 | -1.7 (5.7) | -2.0 (4.5)
  Week 6: number analyzed (Participants) | 75 | 73
  Week 6 | -0.8 (5.8) | -1.7 (5.5)
  Week 8: number analyzed (Participants) | 70 | 66
  Week 8 | -1.4 (5.3) | -3.2 (5.9)
  Week 10: number analyzed (Participants) | 65 | 64
  Week 10 | -1.5 (6.3) | -2.8 (6.7)
  Week 12: number analyzed (Participants) | 64 | 62
  Week 12 | -2.0 (5.9) | -3.0 (6.7)

9. Secondary Outcome: Change From Baseline Beck Anxiety Index (BAI) Total Score
Description: BAI is a 21-item participant-completed questionnaire designed to assess the characteristics of anxiety. Each item is rated on a 4-point scale (0= not present; 3= present in the extreme). Total scores range from 0 to 63. Higher total scores indicate greater severity of anxiety symptoms.
Time Frame: Baseline, Weeks 6 and 12
Population: All randomized participants who received at least one dose of study drug and had BAI assessed at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 75 | 73
units on a scale
  Week 6 | -1.9 (6.6) | -2.3 (7.2)
  Week 12: number analyzed (Participants) | 63 | 62
  Week 12 | -1.3 (6.7) | -2.0 (6.8)

10. Secondary Outcome: Change From Baseline in Plasma Gamma-Glutamyl Transferase (GGT)
Time Frame: Baseline, Weeks 1 and 2 and 3 and 4 and 6 and 8 and 10 and 12
Population: All randomized participants who received at least one dose of study drug and had GGT assessed at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 91 | 89
units per liter (U/L)
  Week 1 | -5.4 (18.8) | -1.3 (9.4)
  Week 2: number analyzed (Participants) | 86 | 83
  Week 2 | -6.6 (20.2) | -2.1 (12.9)
  Week 3: number analyzed (Participants) | 81 | 76
  Week 3 | -9.7 (26.1) | -3.7 (13.7)
  Week 4: number analyzed (Participants) | 78 | 76
  Week 4 | -8.0 (27.3) | -3.0 (14.2)
  Week 6: number analyzed (Participants) | 74 | 72
  Week 6 | -10.9 (33.4) | -4.1 (17.8)
  Week 8: number analyzed (Participants) | 70 | 63
  Week 8 | -10.9 (36.2) | -3.4 (20.6)
  Week 10: number analyzed (Participants) | 64 | 64
  Week 10 | -12.2 (35.8) | -4.0 (26.4)
  Week 12: number analyzed (Participants) | 62 | 61
  Week 12 | -11.5 (42.6) | -2.1 (20.1)

11. Secondary Outcome: Change From Baseline in Plasma Carbohydrate Deficient Transferrin (CDT)
Description: Carbohydrate Deficient Transferrin is a laboratory test that measures alcohol consumption. Greater levels suggest recent alcohol consumption.
Time Frame: Baseline, Weeks 1 and 2 and 3 and 4 and 6 and 8 and 10 and 12
Population: All randomized participants who received at least one dose of study drug and had CDT assessed at both baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: percent CDT
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 82 | 83
percent CDT
  Week 1 | -0.1 (0.5) | -0.0 (0.7)
  Week 2: number analyzed (Participants) | 79 | 78
  Week 2 | -0.2 (0.7) | -0.1 (0.8)
  Week 3: number analyzed (Participants) | 74 | 74
  Week 3 | -0.1 (0.9) | -0.0 (1.2)
  Week 4: number analyzed (Participants) | 70 | 72
  Week 4 | -0.2 (0.9) | 0.1 (1.5)
  Week 6: number analyzed (Participants) | 66 | 68
  Week 6 | -0.1 (1.2) | 0.2 (1.5)
  Week 8: number analyzed (Participants) | 61 | 58
  Week 8 | -0.0 (1.4) | 0.1 (1.3)
  Week 10: number analyzed (Participants) | 57 | 60
  Week 10 | -0.1 (1.5) | 0.1 (0.8)
  Week 12: number analyzed (Participants) | 57 | 58
  Week 12 | -0.0 (1.2) | 0.1 (0.7)

12. Secondary Outcome: 12 -Item Short-Form Health Survey (SF-12) Scores: Physical Component Summary (PCS)
Description: Short Form 12 (SF-12) is a 12-item assessment used to measure participant's physical wellbeing [physical component score (PCS)] and mental wellbeing [mental component score (MCS)]. The PCS score ranges from 0 (lowest wellbeing) to 100 (highest wellbeing) and is designed to have a mean of 50 and standard deviation (SD) of 10 in the general population.
Time Frame: Baseline and Week 12
Population: All randomized participants who received at least one dose of study drug and had SF-12 assessed at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 92 | 88
units on a scale
  PCS: Baseline | 49.2 (8.7) | 50.2 (8.3)
  PCS: Week 12: number analyzed (Participants) | 63 | 61
  PCS: Week 12 | 53.0 (8.6) | 51.4 (7.5)

13. Secondary Outcome: 12-Item Short-Form Health Survey (SF-12) Scores: Mental Component Summary (MCS)
Description: Short Form 12 (SF-12) is a 12-item assessment used to measure participant's physical wellbeing [physical component score (PCS)] and mental wellbeing [mental component score (MCS)]. The MCS score ranges from 0 (lowest wellbeing) to 100 (highest wellbeing) and is designed to have a mean of 50 and standard deviation (SD) of 10 in the general population.
Time Frame: Baseline and Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 92 | 88
units on a scale
  MCS: Baseline | 45.7 (11.6) | 44.2 (11.2)
  MCS: Week 12 | 48.5 (10.0) | 49.7 (9.6)

ADVERSE EVENTS:
Arm/Group | LY686017 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/91
Other Adverse Events (participants affected / at risk) | 73/92 | 68/91
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY686017 (N=92) | Placebo (N=91)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 9 (9) | 6 (6)
Nausea (Gastrointestinal disorders) | 7 (8) | 14 (17)
Fatigue (General disorders) | 8 (9) | 7 (8)
Irritability (General disorders) | 0 (0) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 14 (14)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (5)
Dizziness (Nervous system disorders) | 7 (7) | 3 (3)
Headache (Nervous system disorders) | 6 (7) | 9 (13)
Somnolence (Nervous system disorders) | 7 (7) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days